CLINICAL TRIAL: NCT01750060
Title: Pharmacokinetic Characterization of the Active, Separated System With PK Controller (Fentanyl Iontophoretic Transdermal System, 40 Mcg Fentanyl Per Activation).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: PK2011-001
Record Dates: First submitted 2012-12-10; First posted 2012-12-17 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Fentanyl; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Fentanyl citrate IV infusion & Naltrexone (Active Comparator): Fentanyl citrate (equivalent to 80 mcg fentanyl)administered over 20 minutes by IV infusion every hour through 23.33 hours. Naltrexone (50 mg) will be administered orally (PO) every 12 hours, beginning 14 hours before the start of fentanyl treatment and ending approximately 11 hours after completion of treatment regimen to antagonize the clinical opioid effects of fentanyl.
  Interventions: Drug: Fentanyl; Drug: Naltrexone
- Fentanyl Study System (170 mcAmps) & Naltrexone (Experimental): Two consecutive 40 mcg fentanyl doses each delivered over 10 minutes by the Study System (170 mcAmps) every hour through 23.33 hours. Naltrexone (50 mg) will be administered orally (PO) every 12 hours, beginning 14 hours before the start of fentanyl treatment and ending approximately 11 hours after completion of treatment regimen to antagonize the clinical opioid effects of fentanyl.
  Interventions: Drug: Fentanyl; Drug: Naltrexone
- Fentanyl, Study System (140 mcAmp) & Naltrexone (Experimental): Two consecutive 35 mcg fentanyl doses, each delivered over 10 minutes by the Study System (140 mcAmp) every hour through 23.33 hours. Naltrexone (50 mg) will be administered orally (PO) every 12 hours, beginning 14 hours before the start of fentanyl treatment and ending approximately 11 hours after completion of treatment regimen to antagonize the clinical opioid effects of fentanyl.
  Interventions: Drug: Fentanyl; Drug: Naltrexone
- Fentanyl, Study System (200 mcAmp) & Naltrexone (Experimental): Two consecutive 50 mcg fentanyl doses, each delivered over 10 minutes by the Study System (200 mcAmp) every hour through 23.33 hours. Naltrexone (50 mg) will be administered orally (PO) every 12 hours, beginning 14 hours before the start of fentanyl treatment and ending approximately 11 hours after completion of treatment regimen to antagonize the clinical opioid effects of fentanyl.
  Interventions: Drug: Fentanyl; Drug: Naltrexone
- Fentanyl, Study System (230 mcAmp) & Naltrexone (Experimental): Two consecutive 54 mcg fentanyl doses, each delivered over 10 minutes by the Study System (230 mcAmp) every hour through 23.33 hours. Naltrexone (50 mg) will be administered orally (PO) every 12 hours, beginning 14 hours before the start of fentanyl treatment and ending approximately 11 hours after completion of treatment regimen to antagonize the clinical opioid effects of fentanyl.
  Interventions: Drug: Fentanyl; Drug: Naltrexone

INTERVENTIONS:
Drug: Fentanyl
Drug: Naltrexone

SUMMARY:
"This study is a single-center, randomized, open-label, 3-period, 5-treatment, 6-sequence design. A total of 54 eligible subjects will receive three total treatments; one with intravenous (IV) infusion and two with the Study System. Each subject will be randomly assigned to receive a treatment sequence consisting of Treatment A (IV fentanyl citrate), Study System Treatment B (170 mcAmp), and one of three additional Study System treatments (140 mcAmp or 200 mcAmp or 230 mcAmp) "

DETAILED DESCRIPTION:
"The Study System is a single-use system that consists of two parts: a Drug Unit containing 10.8 mg fentanyl hydrochloride, and a Controller that supplies the dosing current. The two parts are packaged separately and assembled immediately prior to use. The Study System will be applied to the upper, outer arm of each subject. Fentanyl will be delivered from the Study System via transdermal iontophoresis using a current of 170 mcAmp (Treatment B), 140 mcAmp (Treatment C), 200 mcAmp (Treatment D), or 230 mcAmp (Treatment E). Each subject will be randomly assigned to a treatment sequence consisting of Treatment A (IV fentanyl citrate), Study System Treatment B (170 mcAmp), and one of three additional Study System treatments consisting of Treatment C (140 mcAmp), Treatment D (200 mcAmp), or Treatment E (230 mcAmp). Each subject will therefore receive a total of three treatments (A and B and either C, D, or E).

The specific treatments are outlined in detail below:

* Treatment A: Fentanyl citrate (equivalent to 80 mcg fentanyl) administered over 20 minutes by IV infusion every hour through 23.33 hours.
* Treatment B: Two consecutive 40 mcg fentanyl doses each delivered over 10 minutes by the Study System (170 mcAmp) every hour through 23.33 hours.
* Treatment C: Two consecutive 35 mcg fentanyl doses, each delivered over 10 minutes by the Study System (140 mcAmp) every hour through 23.33 hours.
* Treatment D: Two consecutive 50 mcg fentanyl doses, each delivered over 10 minutes by the Study System (200 mcAmp) every hour through 23.33 hours.
* Treatment E: Two consecutive 54 mcg fentanyl doses, each delivered over 10 minutes by the Study System (230 mcAmp) every hour through 23.33 hours.

Naltrexone (50 mg) will be administered orally (PO) every 12 hours, beginning 14 hours before the start of each fentanyl treatment and ending approximately 11 hours after completion of each treatment "

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide written informed consent to participate in the study and document their understanding that they are free to withdraw from the study at any time.
2. Subjects must be healthy volunteers with no clinically relevant abnormalities, as determined by medical history, physical examination, blood chemistry, complete blood count, routine urinalysis (a microscopic urine analysis will be performed at the Investigator's discretion if the macroscopic analysis is abnormal), and electrocardiogram (ECG). Prior medical history, physical examination, and physical and laboratory findings will be reviewed and repeated as deemed appropriate by the supervising physician.
3. Subjects must be male or female volunteers, between ages 18 to 45 years, inclusive.
4. Subjects must have a Body Mass Index (BMI = weight [kg]/height2 [m2] of 18 to 28 kg/m2, inclusive.
5. Subjects must have an average blood pressure from three separate readings in the range of 100 to 139 mm Hg systolic (inclusive) and 50 and 89 mm Hg diastolic (inclusive) after sitting for 5 minutes before and between readings.
6. Subjects must have negative urine drug test results (for drugs of abuse) in each urine sample collected at the time of fentanyl dosing in each treatment period. Each urine sample will be tested for the presence of cannabinoids, amphetamines, barbiturates, benzodiazepines, cocaine, and opiates.
7. Subjects must have a negative alcohol test within the 24 hours before the start of fentanyl dosing in each treatment period.
8. Subjects must provide consent to use a medically acceptable method of contraception throughout the entire duration of the study and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and/or female partner include birth control pills, diaphragm with spermicide, intrauterine device (IUD), condom with spermicide, vaginal spermicidal suppository, surgical sterilization (6 months post-surgery), post-menopausal (not experienced a menstrual period for a minimum of 2 years), and progestin implant or injection (used consistently for the 3 months prior to study dosing).

Exclusion Criteria:

1. Subjects who are pregnant or plan to become pregnant during the time of their participation in this study
2. Subjects with clinically significant medical problems that, in the opinion of the supervising principal investigator, place the subject at undue risk of AEs. These conditions can include, but are not limited to, dermatologic, psychiatric, respiratory, cardiovascular, hepatic, renal, gastrointestinal, hematological, genitourinary, gynecologic, neurologic, or endocrine or other organ abnormality or pathology.
3. Subjects with evidence of orthostatic hypotension (e.g., supine-to-standing blood pressure decrease of ≥ 20 mm Hg systolic or ≥ 10 mm Hg diastolic AND ≥ 20 beats per minute (bpm) increase in heart rate after standing for 3 minutes) or with any reported symptoms of lightheadedness, dizziness, or fainting upon standing.
4. Subjects with resting heart rate < 50 or > 100 beats per minute.
5. Subjects with a history of chronic obstructive pulmonary disease (COPD) or any other lung disease (e.g., sleep apnea,asthma) that could cause CO2 retention beyond normal.
6. Subjects with oxygen saturation < 97% on room air.
7. Subjects with active systemic skin disease or with active local skin disease, such as but not limited to, sunburn, psoriasis, or atopic dermatitis, which would preclude application of the Study System to the upper outer arm.
8. Subjects with a history of significant dermatologic cancers (e.g., melanoma or squamous cell carcinoma). Basal cell carcinomas that were superficial and do not involve the arms are acceptable.
9. Subjects with localized skin pigmentation (e.g., tattoos, sunburn, scars, branding, etc.) or open sores, body piercing, active skin lesions on the upper arms that could interfere with the ability to assess skin site reactions.
10. Subjects with excessive body hair at the intended application site and who refuse hair clipping at the application site
11. Subjects with a known allergy or hypersensitivity to fentanyl or other opioids, naltrexone, naloxone, cetylpyridinium chloride, skin adhesives, tapes, or other transdermal systems
12. Subjects who have reported using:

    * prescription medication (except for sex-hormone replacement or birth control) within 14 days prior to Day 0 of the first treatment period
    * over-the-counter (OTC) medication (except for multivitamin supplements or acetaminophen < 2 g/day) within 3 days prior to Day 0 of the first treatment period
    * alcohol, grapefruit juice, Seville oranges (e.g., marmalade), caffeine, or xanthine-containing products within 48 hours prior to dosing in each fentanyl treatment group
    * daily doses of herbal medication (e.g., Hypericum perforatum [St. John's Wort], Ephedra, Ginkgo, Ginseng, or garlic supplement) within 14 days before Day 0 of the first treatment period
    * prescription or OTC topical medications on the arms, including but not limited to corticosteroids and retinoids, within 28 days
13. Subjects planning to take prescription, OTC, or herbal medications from Day 0 of the first treatment period to the last study assessment with the exception of sex-hormone replacement, birth control, multivitamins, or acetaminophen (< 2 g/day). NOTE: use of topical medications, including antibiotics and corticosteroids, required to treat skin irritation resulting from application of the Study System is allowed.
14. Subjects who have received an investigational drug within the longer of: (a) the past 28 days, or (b) a period of five times the drug's half-life.
15. Subjects with a history or presence of drug or alcohol dependence or abuse.
16. Subjects who smoke > 10 cigarettes, 2 cigars, or 2 tobacco pipes per day within the last 6 months, as determined by medical history and/or subject's verbal report.
17. Subjects who are unable to abstain from smoking during the treatment periods.
18. Subjects who consume alcohol in quantities > 2 alcohol drinks every day, where 1 alcohol drink is defined as 12 ounces of beer, 1 ounce of hard liquor, or 4 ounces of wine.
19. Subjects who exhibit one or more signs or symptoms of opioid withdrawal due to the naloxone challenge test as determined by the Investigator(s).
20. Males with hemoglobin < 12.5 g/dL and females with hemoglobin < 11.5 g/dL.
21. Subjects who have donated blood, experienced a blood loss of > 400 mL within 28 days before dosing, or who plan to donate blood during the study.
22. Subjects who donated plasma within 7 days prior to dosing, or who plan to donate plasma during the study.
23. Subjects who are febrile (temperature > 100.3ºF) at check-in for each treatment period.
24. Subjects who are known to have tested positive for HIV or hepatitis B or hepatitis C.
25. Employees of the investigator or study center, as well as family members of the employees or the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Measure area under the fentanyl concentration-time curve (AUC) | The two-hour period for hours 23-24 for all treatment groups.
  Measure area under the fentanyl concentration-time curve (AUC), one of the five key pharmacokinetic (PK) parameters for the Active, Separated System with PK Controller in the study population.
Measure maximum fentanyl concentration (Cmax) | The two-hour period for hours 23-24 for all treatment groups.
  Measure maximum fentanyl concentration (Cmax), one of the five key pharmacokinetic (PK) parameters for the Active, Separated System with PK Controller in the study population.
Measure time to Cmax (tmax) | The two-hour period for hours 23-24 for all treatment groups.
  Measure time to Cmax (tmax), one of the five key pharmacokinetic (PK) parameters for the Active, Separated System with PK Controller in the study population.
Measure terminal half-life (t½) | The two-hour period for hours 23-24 for all treatment groups.
  Measure terminal half-life (t½), one of the five key pharmacokinetic (PK) parameters for the Active, Separated System with PK Controller in the study population.
Measure the amount of fentanyl absorbed | The two-hour period for hours 23-24 for all treatment groups.
  Measure the amount of fentanyl absorbed, one of the five key pharmacokinetic (PK) parameters for the Active, Separated System with PK Controller in the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Robert I. Cooper, M.D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States